CLINICAL TRIAL: NCT02613507
Title: An Open-label Randomized Multinational Phase 3 Trial of Nivolumab Versus Docetaxel in Previously Treated Subjects With Advanced or Metastatic Non-small Cell Lung Cancer (CheckMate 078: CHECKpoint Pathway and nivoluMAb Clinical Trial Evaluation 078)
Brief Title: Efficacy Study of Nivolumab Compared to Docetaxel in Subjects Previously Treated With Advanced or Metastatic Non Small Cell Lung Cancer
Acronym: CheckMate 078
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-078; 2015-001893-16 (EudraCT Number)
Record Dates: First submitted 2015-11-22; First posted 2015-11-24 (Estimated); Results first posted 2019-02-22 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Nivolumab (Experimental): Nivolumab Intravenous infusion specified dose on specified days
  Interventions: Drug: Nivolumab
- Arm B: Docetaxel (Active Comparator): Docetaxel Intravenous infusion specified dose on specified days
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Nivolumab
  Arms: Arm A: Nivolumab
Drug: Docetaxel
  Arms: Arm B: Docetaxel

SUMMARY:
The purpose of this study is to determine whether Nivolumab improves life expectancy compared to Docetaxel in Subjects with Advanced or Metastatic Non-small Cell Lung Cancer who have failed prior platinum-based doublet chemotherapy.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Disease progression experienced during or after one prior platinum containing doublet chemotherapy
* Stage IIIb/IV or recurrent disease
* Male and Female ≥ 18 years of age
* Measurable disease per RECIST 1.1
* Performance Status ≤ 1

Exclusion Criteria:

* History of Carcinomatous meningitis
* Active Central nervous system (CNS) metastases
* History of auto immune diseases
* Prior treatment with Docetaxel
* Prior treatment with ipilimumab or any drug targeting T-Cell costimulation or checkpoint pathways

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2015-12-11 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2023-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (33):
- China (24):
  - Local Institution - 0051, Beijing, Beijing Municipality
  - Local Institution - 0007, Beijing, Beijing Municipality
  - Local Institution - 0032, Beijing, Beijing Municipality
  - Local Institution - 0026, Beijing, Beijing Municipality
  - Local Institution - 0020, Chongqing, Chongqing Municipality
  - Local Institution - 0015, Fuzhou, Fujian
  - Local Institution - 0003, Guangzhou, Guangdong
  - Local Institution - 0002, Guangzhou, Guangdong
  - Local Institution - 0024, Zhengzhou, Henan
  - Local Institution - 0023, Changsha, Hunan
  - Local Institution - 0012, Changsha, Hunan
  - Local Institution - 0034, Nanjing, Jiangsu
  - Local Institution - 0006, Changchun, Jilin
  - Local Institution - 0022, Changchun, Jilin
  - Local Institution - 0017, Shanghai, Shanghai Municipality
  - Local Institution - 0025, Shanghai, Shanghai Municipality
  - Local Institution - 0011, Chengdu, Sichuan
  - Local Institution - 0008, Hangzhou, Zhejiang
  - Local Institution - 0009, Hangzhou, Zhejiang
  - Local Institution - 0010, Hangzhou, Zhejiang
  - Local Institution - 0031, Beijing
  - Local Institution - 0029, Beijing
  - Local Institution - 0014, Shanghai
  - Local Institution - 0028, Shanghai
- Local Institution - 0049, Hong Kong, Hong Kong
- Russia (6):
  - Local Institution - 0039, Chelyabinsk
  - Local Institution - 0052, Moscow
  - Local Institution - 0046, Moscow
  - Local Institution - 0042, Saint Petersburg
  - Local Institution - 0040, Saint Petersburg
  - Local Institution - 0041, Saint Petersburg
- Singapore (2):
  - Local Institution - 0048, Singapore
  - Local Institution - 0037, Singapore

REFERENCES:
- [Derived] Hu S, Tang Z, Harrison JP, Hertel N, Penrod JR, May JR, Juarez-Garcia A, Holdgate O. Economic Evaluation of Nivolumab Versus Docetaxel for the Treatment of Advanced Squamous and Non-squamous Non-small Cell Lung Cancer After Prior Chemotherapy in China. Pharmacoecon Open. 2023 Mar;7(2):273-284. doi: 10.1007/s41669-022-00383-x. Epub 2023 Mar 10. PMID 36897427
- [Derived] Wu YL, Lu S, Cheng Y, Zhou C, Wang J, Mok T, Zhang L, Tu HY, Wu L, Feng J, Zhang Y, Luft AV, Zhou J, Ma Z, Lu Y, Hu C, Shi Y, Baudelet C, Cai J, Chang J. Nivolumab Versus Docetaxel in a Predominantly Chinese Patient Population With Previously Treated Advanced NSCLC: CheckMate 078 Randomized Phase III Clinical Trial. J Thorac Oncol. 2019 May;14(5):867-875. doi: 10.1016/j.jtho.2019.01.006. Epub 2019 Jan 17. PMID 30659987
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT02613507.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Nivolumab: 3 mg/kg every 2 weeks until disease progression or unacceptable toxicity
- Docetaxel: 75 mg/m² every 3 weeks until disease progression or unacceptable toxicity
Period: Pre-Treamtent
Arm/Group | Nivolumab | Docetaxel
Started (Randomized) | 338 | 166
Completed (Received Treatment) | 337 | 156
Not Completed | 1 | 10
Not completed — Participant request to discontinue study treatment | 0 | 5
Not completed — Participant withdrew consent | 0 | 4
Not completed — Participant no longer meets study criteria | 1 | 1
Period: Treatment
Arm/Group | Nivolumab | Docetaxel
Started (Treated) | 337 | 156
Crossover to Nivolumab (Participants from the Docetaxel arm who changed treatment arms to receive Nivolumab) | 0 | 9
Completed (Continuing in the study) | 0 | 0
Not Completed | 337 | 156
Not completed — Not reported | 3 | 0
Not completed — Other reasons | 8 | 0
Not completed — Participant no longer meets criteria | 3 | 0
Not completed — Maximum clinical benefit | 5 | 10
Not completed — Lost to Follow-up | 1 | 0
Not completed — Participant withdrew consent | 0 | 2
Not completed — Participant request to discontinue study treatment | 13 | 17
Not completed — Adverse event unrelated to study drug | 20 | 3
Not completed — Death | 2 | 0
Not completed — Study drug toxicity | 19 | 14
Not completed — Disease progression | 263 | 110

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab | Docetaxel | Total
Number analyzed (Participants) | 338 | 166 | 504
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.1 (9.07) | 59.3 (8.13) | 59.1 (8.77)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 263 | 134 | 397
  Female | 75 | 32 | 107
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 30 | 15 | 45
  Chinese | 306 | 151 | 457
  Asian Other | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Median Overall Survival
Description: OS was defined as the time between the date of randomization and the date of death. For subjects without documentation of death, OS was censored on the last date the subject was known to be alive
Time Frame: From randomization to the date of death or date participant was last known to be alive (assessed from December 2015 to Oct 2017 approximately 22 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab | Docetaxel
Number analyzed (Participants) | 338 | 166
Months | 11.99 [10.35 to 14.00] | 9.63 [7.62 to 11.24]
Statistical Analysis 1: Comparison: Nivolumab vs Docetaxel; Test type: Superiority; p = 0.0006, Stratified weighted Log-Rank — The boundary for statistical significance requires the p-value to be less than 0.0231; Stratified weighted using G [rho=0, gamma=1] Fleming and Harrington
Statistical Analysis 2: Comparison: Nivolumab vs Docetaxel; Test type: Superiority; Stratified Cox Proportional Hazard Model; Hazard Ratio (HR) = 0.68, 97.7% CI 2-sided [0.52 to 0.90]
Statistical Analysis 3: Comparison: Nivolumab vs Docetaxel; Test type: Superiority; p = 0.0017, Log Rank; regular stratified log-rank test p-value

2. Primary Outcome: Overall Survival Rate
Description: OS was defined as the time between the date of randomization and the date of death. For subjects without documentation of death, OS was censored on the last date the subject was known to be alive. Rates provided are Kaplan-Meier estimates.
Time Frame: From first dose to the date of death or date participant was last known to be alive (assessed from December 2015 to Oct 2017 approximately 22 months)
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Nivolumab | Docetaxel
Number analyzed (Participants) | 338 | 166
percentage
  Rate at 6 months | 72.4 [67.3 to 76.9] | 64.8 [56.8 to 71.6]
  Rate at 12 months | 49.7 [44.1 to 55.0] | 38.8 [31.1 to 46.5]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: Investigator assessed ORR was defined as the number of participants whose best objective response (BOR) was a confirmed complete response (CR) or confirmed partial response (PR), as determined by the investigator, divided by the number of randomized participants.
  CR= Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR= At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From date of first dose up to partial or complete response (up to approximately 90 months)
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab | Docetaxel
Number analyzed (Participants) | 338 | 166
Percentage of participants
  All randomized participants | 17.5 [13.6 to 21.9] | 4.2 [1.7 to 8.5]
  Squamous NSCLC: number analyzed (Participants) | 133 | 67
  Squamous NSCLC | 21.1 [14.5 to 29.0] | 1.5 [0.0 to 8.0]
  Non-Squamous NSCLC: number analyzed (Participants) | 205 | 99
  Non-Squamous NSCLC | 15.1 [10.5 to 20.8] | 6.1 [2.3 to 12.7]
  PD-L1 >= 1%: number analyzed (Participants) | 168 | 84
  PD-L1 >= 1% | 17.3 [11.9 to 23.8] | 6.0 [2.0 to 13.3]
  PD-L1 < 1%: number analyzed (Participants) | 138 | 67
  PD-L1 < 1% | 18.1 [12.1 to 25.6] | 3.0 [0.4 to 10.4]
  PD-L1 Non-quantifiable: number analyzed (Participants) | 32 | 15
  PD-L1 Non-quantifiable | 15.6 [5.3 to 32.8] | NA [0.0 to 21.8] — NA= Number not calculated due to insufficient number of events.
  Chinese: number analyzed (Participants) | 302 | 149
  Chinese | 17.2 [13.1 to 22.0] | 3.4 [1.1 to 7.7]
  Non-Chinese: number analyzed (Participants) | 36 | 17
  Non-Chinese | 19.4 [8.2 to 36.0] | 11.8 [1.5 to 36.4]

4. Secondary Outcome: Overall Survival (OS) in Subpopulations
Description: OS was defined as the time between the date of randomization and the date of death. For participants without documentation of death, OS was censored on the last date the participant was known to be alive. Test stratified by histology (SQ vs NSQ), PD-L1 status at 1% expression level (positive vs negative/unevaluable).
Time Frame: From randomization to the date of death or date participant was last known to be alive (up to approximately 90 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab | Docetaxel
Number analyzed (Participants) | 338 | 166
Months
  Greater than/equal to 1% PD-L1 expression: number analyzed (Participants) | 168 | 84
  Greater than/equal to 1% PD-L1 expression | 11.99 [10.18 to 14.55] | 7.89 [5.32 to 9.63]
  Less than 1% PD-L1 expression: number analyzed (Participants) | 138 | 67
  Less than 1% PD-L1 expression | 11.37 [8.84 to 15.34] | 10.25 [7.62 to 13.83]
  Non-quantifiable PD-L1 Expression: number analyzed (Participants) | 32 | 15
  Non-quantifiable PD-L1 Expression | 15.57 [7.10 to 20.44] | 16.30 [5.45 to 26.12]
  Histologically Squamous: number analyzed (Participants) | 133 | 67
  Histologically Squamous | 11.70 [8.87 to 14.00] | 7.89 [5.88 to 11.20]
  Histologically Non-squamous: number analyzed (Participants) | 205 | 99
  Histologically Non-squamous | 11.86 [9.40 to 15.34] | 10.22 [7.82 to 13.11]
  Chinese participants: number analyzed (Participants) | 302 | 149
  Chinese participants | 11.76 [10.18 to 13.80] | 8.57 [6.93 to 10.25]
  Non-Chinese participants: number analyzed (Participants) | 36 | 17
  Non-Chinese participants | 12.98 [8.61 to 20.57] | 16.30 [5.16 to 21.36]

5. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from randomization to the date of the first documented tumor progression as determined by investigators per RECIST 1.1, or death due to any cause. Clinical deterioration in the absence of unequivocal evidence of progression was not considered progression for purposes of determining PFS. Participants who died without a reported prior progression were considered to have progressed on the date of their death. Participants who did not have disease progression or die were censored on the date of their last evaluable tumor assessment. Participants who did not have any on study tumor assessments and did not die were censored at the randomization date. Participants who started any subsequent anti-cancer therapy (including on-treatment palliative RT of non-target bone lesions, skin lesions or CNS lesions) without a prior reported progression were censored at the last evaluable tumor assessment prior to or on initiation of the subsequent anti-cancer therapy.
Time Frame: From the time of randomization to the date of the first documented tumor progression or death due to any cause (up to approximately 90 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab | Docetaxel
Number analyzed (Participants) | 338 | 166
Months
  All randomized participants | 2.79 [2.37 to 3.65] | 2.76 [1.81 to 3.02]
  Histologically Squamous: number analyzed (Participants) | 133 | 67
  Histologically Squamous | 2.92 [2.37 to 4.17] | 2.66 [1.45 to 2.92]
  Histologically Non-Squamous: number analyzed (Participants) | 205 | 99
  Histologically Non-Squamous | 2.60 [1.54 to 3.91] | 2.83 [1.64 to 4.11]
  PD-L1 >= 1%: number analyzed (Participants) | 168 | 84
  PD-L1 >= 1% | 2.76 [1.68 to 4.01] | 2.56 [1.48 to 2.99]
  PD-L1 < 1%: number analyzed (Participants) | 138 | 67
  PD-L1 < 1% | 2.86 [1.71 to 4.11] | 2.78 [1.41 to 4.24]
  PD-L1 Non-quantifiable: number analyzed (Participants) | 32 | 15
  PD-L1 Non-quantifiable | 2.00 [1.35 to 5.55] | 4.07 [1.41 to 6.93]
  Chinese participants: number analyzed (Participants) | 302 | 149
  Chinese participants | 2.76 [2.04 to 3.35] | 2.69 [1.54 to 2.83]
  Non-Chinese participants: number analyzed (Participants) | 36 | 17
  Non-Chinese participants | 3.50 [1.48 to 9.40] | 8.48 [2.23 to 16.30]

6. Secondary Outcome: Progression Free Survival Rate
Description: Clinical deterioration in the absence of unequivocal evidence of progression (per RECIST 1.1) is not considered progression for purposes of determining PFS. Participants who die without a reported prior progression will be considered to have progressed on the date of their death. Participants who did not have disease progression or die will be censored on the date of their last evaluable tumor assessment. Participants who did not have any on study tumor assessments and did not die will be censored at the randomization date. Participants who started any subsequent anti-cancer therapy without a prior reported progression will be censored at the last evaluable tumor assessment prior to or on initiation of the subsequent anti-cancer therapy. Six month progression-free survival rate as estimated using the Kaplan-Meier method
Time Frame: From the time of randomization up to 6 months
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Nivolumab | Docetaxel
Number analyzed (Participants) | 338 | 166
Percentage | 29.3 [24.4 to 34.3] | 24.8 [18.0 to 32.1]

7. Secondary Outcome: Time to Treatment Failure (TTF)
Description: TTF was defined as the minimum of the time from randomization to disease progression (per RECIST 1.1 or clinical), death or last dose date if a participant discontinued from treatment for any reasons other than "maximum clinical benefit" and "administrative reasons by sponsor". TTF was considered as event at the randomization date for participants who were randomized but not treated. TTF was censored at the last dose date for participants who discontinued treatment due to "maximum clinical benefit" or "administrative reasons by sponsor". TTF was censored at the last dose date for participants who continued on treatment without progression or death.
  This outcome measure was prespecified in the protocol to only be evaluated through the first Interim Analysis, which occurred in June 2017.
Time Frame: From randomization up to disease progression, death, or last dose (up to approximately 17 months)
Population: All randomized participants with at least 8 months of follow-up at the time of TTF analysis. The clinical database cutoff date will occur when the first approximately 380 randomized participants will have at least 8-month of follow-up.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab | Docetaxel
Number analyzed (Participants) | 258 | 131
Months | 2.60 [1.81 to 2.92] | 1.51 [1.41 to 2.23]

8. Secondary Outcome: Number of Participants Experiencing Treatment-Related Adverse Events (AEs)
Description: A treatment-related Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study treatment and is determined to be associated with the study treatment. Adverse events are graded on a scale from 1 to 5, with Grade 1 being mild and asymptomatic; Grade 2 is moderate requiring minimal, local or noninvasive intervention; Grade 3 is severe or medically significant but not immediately life-threatening; Grade 4 events are usually severe enough to require hospitalization; Grade 5 events are fatal.
Time Frame: From first dose up to 100 days after last dose (up to 93 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab | Docetaxel
Number analyzed (Participants) | 337 | 156
Participants | 220 | 131

9. Secondary Outcome: Number of Participants Experiencing Treatment-Related Serious Adverse Events (SAEs)
Description: A treatment-related Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening (defined as an event in which the participant was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe), requires inpatient hospitalization or causes prolongation of existing hospitalization and is determined to be associated with the study treatment.
Time Frame: From first dose up to 100 days after last dose (up to 93 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab | Docetaxel
Number analyzed (Participants) | 337 | 156
Participants | 34 | 25

10. Secondary Outcome: Disease Related Symptom Deterioration Rate by Week 12 and Week 24
Description: Disease-Related Symptom Deterioration Rate is the percentage of participants with >=10 points increase from baseline in Average Symptom Burden Index (ASBI) score at any time between randomization and the timepoints. The Lung Cancer Symptom Scale (LCSS) measures 6 items (loss of appetite, fatigue, coughing, shortness of breath, hemoptysis, pain) and 3 symptom burden items (disease-related functional limitations, quality of life) with responses captured using a 100mm visual analog scale (VAS). Scores range from 0 (highest quality of life) to 100 (worst quality of life) and is derived by dividing the length of the line drawn from the lowest possible response to the patient's response by the length of the VAS and multiplying the result by 100. An ASBI score can be derived as the mean of scores for the 6 symptom-related items with a clinically meaningful change in ASBI score being 10 points and a meaningful deterioration in symptoms is a mean post-baseline score change >= 10 points.
Time Frame: At Week 12 and Week 24
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab | Docetaxel
Number analyzed (Participants) | 338 | 166
Percentage of participants
  Week 12 | 29.9 [25.0 to 35.1] | 40.4 [32.8 to 48.2]
  Week 24 | 34.6 [29.6 to 40.0] | 42.2 [34.6 to 50.1]

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their randomization to study completion, (up to approximately 95 months). SAEs and Other AEs were assessed from first dose to 100 days following last dose (up to approximately 93 months)
Groups:
- Cross-over Nivolumab: Participants from the Docetaxel arm who changed treatment arms to receive Nivolumab 3 mg/kg every 2 weeks until disease progression or unacceptable toxicity
Arm/Group | Nivolumab | Docetaxel | Cross-over Nivolumab
All-Cause Mortality (participants affected / at risk) | 294/337 | 146/156 | 8/9
Serious Adverse Events (participants affected / at risk) | 183/337 | 73/156 | 4/9
Other Adverse Events (participants affected / at risk) | 318/337 | 146/156 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab (N=337) | Docetaxel (N=156) | Cross-over Nivolumab (N=9)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 6 | 0
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Myelosuppression (Blood and lymphatic system disorders) | 1 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute left ventricular failure (Cardiac disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Malignant ascites (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0
Death (General disorders) | 5 | 1 | 0
Disease progression (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 2 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Pain (General disorders) | 2 | 0 | 0
Pyrexia (General disorders) | 2 | 1 | 0
Sudden death (General disorders) | 0 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 4 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 1 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Lung abscess (Infections and infestations) | 1 | 0 | 0
Perinephritis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 37 | 8 | 0
Pneumonia aspiration (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0
Tuberculosis (Infections and infestations) | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 4 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Amylase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0
Body temperature increased (Investigations) | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0
Lipase increased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 4 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0
White blood cell count decreased (Investigations) | 2 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 91 | 36 | 2
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 9 | 0 | 0
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 9 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin oedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab (N=337) | Docetaxel (N=156) | Cross-over Nivolumab (N=9)
Anaemia (Blood and lymphatic system disorders) | 117 | 66 | 4
Leukopenia (Blood and lymphatic system disorders) | 31 | 32 | 0
Myelosuppression (Blood and lymphatic system disorders) | 7 | 11 | 0
Neutropenia (Blood and lymphatic system disorders) | 21 | 31 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 22 | 10 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1 | 1
Palpitations (Cardiac disorders) | 2 | 2 | 1
Hypothyroidism (Endocrine disorders) | 18 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 16 | 6 | 1
Constipation (Gastrointestinal disorders) | 47 | 17 | 4
Diarrhoea (Gastrointestinal disorders) | 36 | 14 | 2
Faeces hard (Gastrointestinal disorders) | 2 | 0 | 1
Gastritis (Gastrointestinal disorders) | 2 | 0 | 1
Nausea (Gastrointestinal disorders) | 38 | 17 | 3
Toothache (Gastrointestinal disorders) | 10 | 1 | 1
Vomiting (Gastrointestinal disorders) | 27 | 18 | 0
Asthenia (General disorders) | 26 | 13 | 0
Chest discomfort (General disorders) | 15 | 8 | 1
Chest pain (General disorders) | 5 | 1 | 1
Fatigue (General disorders) | 105 | 62 | 0
Malaise (General disorders) | 6 | 2 | 1
Non-cardiac chest pain (General disorders) | 42 | 9 | 1
Oedema peripheral (General disorders) | 13 | 9 | 0
Pain (General disorders) | 34 | 15 | 1
Pyrexia (General disorders) | 59 | 28 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 17 | 3 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 3 | 0 | 2
Pneumonia (Infections and infestations) | 34 | 14 | 2
Upper respiratory tract infection (Infections and infestations) | 38 | 8 | 1
Alanine aminotransferase increased (Investigations) | 66 | 18 | 1
Amylase increased (Investigations) | 38 | 3 | 0
Aspartate aminotransferase increased (Investigations) | 63 | 11 | 1
Bilirubin conjugated increased (Investigations) | 14 | 3 | 1
Blood albumin decreased (Investigations) | 12 | 9 | 0
Blood alkaline phosphatase increased (Investigations) | 35 | 2 | 0
Blood creatine phosphokinase MB increased (Investigations) | 2 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 4 | 0 | 1
Blood creatinine increased (Investigations) | 27 | 7 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 6 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 40 | 6 | 0
Haemoglobin decreased (Investigations) | 9 | 15 | 0
Lipase increased (Investigations) | 37 | 2 | 0
Lymphocyte count decreased (Investigations) | 9 | 4 | 1
Neutrophil count decreased (Investigations) | 22 | 32 | 1
Platelet count decreased (Investigations) | 10 | 10 | 1
Weight decreased (Investigations) | 59 | 5 | 3
Weight increased (Investigations) | 23 | 1 | 0
White blood cell count decreased (Investigations) | 32 | 42 | 1
Decreased appetite (Metabolism and nutrition disorders) | 106 | 52 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 28 | 5 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 14 | 3 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 26 | 16 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 12 | 9 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 23 | 6 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 25 | 8 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 55 | 10 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 9 | 2 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 31 | 14 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 31 | 7 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 35 | 9 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 11 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 13 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Diplegia (Nervous system disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 22 | 7 | 0
Headache (Nervous system disorders) | 18 | 3 | 1
Hypoaesthesia (Nervous system disorders) | 16 | 10 | 0
Neuropathy peripheral (Nervous system disorders) | 3 | 8 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 24 | 14 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 4 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 17 | 10 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 104 | 43 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 63 | 27 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 50 | 26 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 45 | 16 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 19 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 12 | 37 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 39 | 5 | 1
Rash (Skin and subcutaneous tissue disorders) | 54 | 9 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication

DOCUMENTS (2):
  • Study Protocol (2017-12-13): https://cdn.clinicaltrials.gov/large-docs/07/NCT02613507/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-02): https://cdn.clinicaltrials.gov/large-docs/07/NCT02613507/SAP_001.pdf